CLINICAL TRIAL: NCT06156917
Title: Evaluation of Autonomic, Imaging and Genetic Markers for Parkinson-related Dementia : Longitudinal Assessment of a PD Cohort.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: AIG/PD CARIPLO grant 2014-0832
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: diagnostic accuracy — Aims of the present project are: to investigate the relationship between incident PD dementia and multimodal parameters as cardiovascular autonomic dysfunction, altered cerebral glucose metabolism, and genetic biomarkers; development of an algorithm predictive for PD-related dementia, combining the rele- vant multidimensional parameters under study; longitudinal follow-up of clinical and cognitive status in PD patients with and without dementia along four years.

SUMMARY:
Neuropathologically, Parkinson disease (PD) is characterized by the accumulation of intra-neuronal protein aggregates (Lewy bodies and Lewy neurites). It is believed that altered rt-synuclein protein handling plays a key role in the etiopathogenesis of PD, because it is the principal component of Lewy pathology. Recent evidence now suggests the possibility that a-synuclein is a prion-like protein and that PD is a prion-like disease. Some studies have suggested that environmental toxins promote the release of a-synuclein by enter- ic neurons and that released enteric a-synuclein is taken up by presynaptic sympathetic neurites and retro- gradely transported to the soma, where it accumulates, thus mediating the progression of PD pathology. These data indicate the precocity of autonomic nervous system involvement with reference to further spread of a-synuclein pathology. We have evidence from a previous study that the vagal preganglionic pro- jections to the gut express a-synuclein, thus providing a candidate a-synuclein-expressing pathway for the retrograde transport of pathogens to the central nervous system. Cardiovascular autonomic dysfunction explores the reactivity of sympathetic and parasympathetic pathways to a predefined set of tests, allowing to quantify the degree of dysfunction in each of the two components of the autonomic nervous system.

Mutations in the GBA gene influence the risk for dementia in PD 21; this effect of GBA is not synergistic with that of increasing age. Heterozygous GBA mutations are considered an important risk factor for PD and dementia, possibly causing a wider protein accumulation in the brain. In vitro models of alpha-synuclein aggregation have provided evidence for co-localization with mutant GBA . It has been proposed that a gain of function mechanism operates in patients with PD carrying GBA gene mutations, whereby mutant G8A promotes alpha-synuclein aggregation, accelerating Lewy body formation and neuronal loss.

Each of the selected variables provides a unique window to ascertain the association between PD patho- physiology and the risk of related dementia. Our hypothesis is that PD patients who develop incident dementia will have a number of statistically different abnormalities that will be evidenced as individual predictors and will also be assembled into a predictive algorithm. This project addresses a key issue in Parkinson disease, a progressive neurodegenerative condition, related to the assessment of variables associated to the development of dementia. The project is focused on dementia as a significant and important clinical milestone that constitutes the main cause of non-reversible functional impairment in PD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "clinically established PD" based on the MDS clinical diagnostic criteria.

Age at disease onset will be between 40 and 70.

Exclusion Criteria:

* severe autonomic dysfunction (as defined in red flag 5a and 5b) will be an exclusion criterion Previous deep brain stimulation is an exclusion criterion.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This project provides the opportunity to collect and characterize a large cohort of PD patients to be studied prospectively.
  We will evaluate whether dlfferences In the measured variables exist between patients who will develop dementia (primary endpoint) within the observatlon time frame and those who will remain free from cognitive impairment at follow-up. We will compare PD patients who reach this endpoint before 10 years from disease onset to those who by that tlme remain cognitively preserved.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
correlation of dysautonomia with incident dementia associated to PD | 2 years
  .At the end of the study, the patients will be divided in two groups: demented and non-demented. Dysauto- nomia measures wili be based on autonomic testing and MIBG scintigraphy.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No